CLINICAL TRIAL: NCT03362021
Title: Comparison of Two Different Sedation Protocol During Transvaginal Oocyte Retrieval: Effects on Propofol Consumption
Brief Title: Comparison of Two Different Sedation Protocols During Transvaginal Oocyte Retrieval
Status: Terminated | Type: Observational
Why Stopped: Primary investigator transferred in another hospital; ongoing pandemic;
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Associate Professor of Anesthesiology, Attikon Hospital
Other Study IDs: TORDEX
Record Dates: First submitted 2017-11-05; First posted 2017-12-05 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Infertility
Keywords: transvaginal oocyte retrieval; sedation; dexmedetomidine; fentanyl; remifentanil; midazolam
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DEX: Sedation with dexmedetomidine (solution 4 γ/ml) continuously infused at a dose of 1 γ/kg/ and fentanyl 100γ iv. Dexmedetomidine infusion will start 10 min before the start of transvaginal oocyte retrieval and will stop at the end of the procedure.
  Interventions: Procedure: transvaginal oocyte retrieval
- MZM: Sedation with remifentanil (solution 50γ/ml) continuously infused at a dose of 0.2 γ/kg/min and midazolam 1 mg iv. Remifentanil infusion will start 10 min before the start of transvaginal oocyte retrieval and will stop at the end of the procedure.
  Interventions: Procedure: transvaginal oocyte retrieval

INTERVENTIONS:
Procedure: transvaginal oocyte retrieval — sedation for oocyte retrieval

SUMMARY:
The effects of two different sedation protocols during transvaginal oocyte retrieval will be investigated on propofol consumption as a rescue sedative and on IVF success. One group will receive dexmedetomidine and fentanyl while the other will receive midazolam and remifentanil.

DETAILED DESCRIPTION:
Women will be consecutively allocated into one of the following two groups using a 1:1 ratio in order to avoid any potential source of bias.

Group DEX: women will receive dexmedetomidine (solution 4 γ/ml) continuously infused at a dose of 1 γ/kg/ and fentanyl 100γ iv. Dexmedetomidine infusion will start 10 min before the start of transvaginal oocyte retrieval and will stop at the end of procedure. At that time point, both total volume (ml) and dose (γ) of dexmedetomidine administered will be recorded.

Group MZM: women will receive remifentanil (solution 50γ/ml) continuously infused at a dose of 0.2 γ/kg/min και midazolam 1 mg iv. Remifentanil infusion will start 10 min before the start of transvaginal oocyte retrieval and will stop at the end of the procedure. At that time point, both total volume (ml) and dose (γ) of remifentanil administered will be recorded.

In both groups, in case of non-co-operation of the woman (e.g. kinetic response), propofol will be given as a bolus rescue dose as follows: the 1st rescue dose will be 1mg/kg while all the next doses will be 0.5 mg/kg. At the end of the procedure, the number of rescue doses and the total rescue dose (mg) of propofol given will be recorded.

Intraoperative monitoring will include ECG, noninvasive blood pressure, SpO2, EtCO2 and depth of sedation using BIS values and ΟΑSS scale. Also, adverse effects such as hypotension, bradycardia, nausea & vomiting, rigidity, airway obstruction, and need for bag-mask ventilation will be recorded. The use of vasoactive drugs will also be reported.

At the end of the procedure, the time and quality of recovery will be assessed using ΟΑSS scale (max score=5), while postoperatively the Post Anesthesia Discharge Scoring System, as well as woman's and gynecologist's (physician) overall satisfaction related to the sedation techniques used, will be recorded.

Regarding the IVF outcome, the following parameters will be recorded: number of oocytes retrieved, the percentage of mature oocytes, embryo quality, percentage of positive pregnancy test, percentage of clinical pregnancy, the percentage of live birth.

ELIGIBILITY:
Inclusion Criteria:

* female patients between 25 and 45 years old that do not meet any of the exclusion criteria

Exclusion Criteria:

* patient refusal, epilepsy, GERD, morbid obesity, drug allergy, ASA class >2, severe hypotension or bradycardia, presence of atrioventricular block, cerebrovascular disease or hepatic dysfunction

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: eligible females scheduled for oocyte retrieval
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
propofol consumption | from the beginning to the end of the transvaginal oocyte retrieval procedure
  difference >30% in propofol consumption

SECONDARY OUTCOMES:
number of oocytes retrieved | up to 3 weeks after starting ovarian stimulation treatment
percentage of mature oocytes | up to 3 weeks after starting ovarian stimulation treatment
fertilization rate | up to 3 weeks after starting ovarian stimulation treatment
embryo quality | up to 4 weeks after starting ovarian stimulation treatment
  Embryo quality for endometrial transfer or cryopreservation will be assessed according to morphological criteria based on the overall blastomere number, size, appearance and degree of fragmentation
positive pregnancy test | up to 3 weeks after transvaginal oocyte retrieval
clinical pregnancy | up to 12 weeks after starting ovarian stimulation treatment
  confirmed presence of an intrauterine sac with fetal heart activity through transvaginal ultrasound scan at seven weeks of gestation, following a positive serum β-hCG test
Live birth | up to 24 weeks after starting ovarian stimulation treatment
  birth of a live fetus after 20 weeks of gestation
BIS score | assessed every 5 minutes during transvaginal oocyte retrieval procedure
  bispectral index score
Observer's Assessment of Alertness/Sedation scale - OAA/S scale | assessed every 5 minutes during transvaginal oocyte retrieval procedure
  used to assess level of sedation during the procedure (5- Responds readily to name spoken in normal tone, 4-Lethargic response to name spoken in normal tone, 3-Responds only after name is called loudly and/or repeatedly, 2-Responds only after mild prodding or shaking, 1-Does not respond to mild prodding or shaking
airway obstruction | during the procedure
  (yes/no)
need to ventilate by mask | during the procedure
  yes/no
presence of muscle rigidity | during the procedure
  yes/no
presence of bradycardia (heart rate less than 50 bpm) | during the procedure
hypotension (mean arterial pressure lower than 65 mmHg) for more than 1' during procedure | during the procedure
dexmedetomidine consumption | from the beginning to the end of the transvaginal oocyte retrieval procedure
  total μg
remifentanil consumption | from the beginning to the end of the transvaginal oocyte retrieval procedure
  total μg
vasoactive drug consumption | from the beginning to the end of the transvaginal oocyte retrieval procedure
patient satisfaction score | end of procedure
  4 point scale (0-poor, 1-good, 2-very good, 3-excellent)
physician satisfaction score | end of procedure
  4 point scale (0-poor, 1-good, 2-very good, 3-excellent)
presence of nausea or vomitus | from end of procedure to discharge from hospital, approximately 4 hours after procedure
  0-none, 1-nausea, 2-vomitus<2, 3 vomitus>2
Post Hospital Discharge Score | from end of procedure to discharge from hospital, approximately 4 hours after procedure
  time required by patient to be able to return at home

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided